CLINICAL TRIAL: NCT03592381
Title: Ridge Expansion by Osseodensification Drilling Compared to Ridge Splitting Technique Simultaneously With Implant Placement in Narrow Alveolar Ridges: A Randomized Controlled Trial
Brief Title: Ridge Expansion by Osseodensification Simultaneously With Implant Placement in Narrow Alveolar Ridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Abdelhamid ElMaghrabi, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422015497758
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Alveolar Ridge Augmentation

STUDY DESIGN:
Intervention Model Description: Double Blinded, Parallel group, Randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ridge expansion by osseodensification (Experimental): Ridge expansion and osteotomy drilling by osseodensification in conjunction with simultaneous implant placement in narrow ridges.
  Interventions: Procedure: Ridge Expansion by ossedensification
- Ridge expansion by ridge splitting (Active Comparator): Ridge expansion by ridge splitting using the piezotome in conjunction with simultaneous implant placement in narrow ridges.
  Interventions: Procedure: ridge expansion by ridge splitting

INTERVENTIONS:
Procedure: Ridge Expansion by ossedensification — Osseodensification is a new concept facilitated by Densah® Burs which are a multi- fluted osteotome like drilling instrumentsThe idea behind the technique is using a non-subtractive drilling mode that preserves bone and increases its density along the osteotomy walls instead of cutting it away (Huwais and Meyer 2015)
  Arms: Ridge expansion by osseodensification
Procedure: ridge expansion by ridge splitting — using the piezotome,Piezoelectric ridge splitting allows exact, clean, and smooth even curved cutting of the bone tissue, with proper visibility.
  Arms: Ridge expansion by ridge splitting

SUMMARY:
Narrow alveolar ridges with a thickness equal or less than 5 mm requires bone augmentation procedures before or at the time of implant placement. (Anitua, Begoña, and Orive 2013) Several surgical techniques have been utilized for the reconstruction of deficient alveolar ridges such as block onlay graft augmentation, guided bone regeneration, distraction osteogenesis , ridge splitting and/or ridge expansion(McAllister and Haghighat 2007). A new bone drilling technique named Osseodensification facilitates horizontal ridge expansion. Studies are needed to validate the effectiveness of osseodensification as a lateral ridge augmentation procedure that aims at increasing the thickness of atrophic ridges, thus maintaining ridge integrity and allowing for implant placement with enhanced stability. The null hypothesis Proposes no difference in the bone width gain following the osseodensification drilling system compared to the ridge splitting technique with simultaneously placed implants in narrow alveolar ridges.

DETAILED DESCRIPTION:
The aim of the study is to evaluate ridge width gain in patients with narrow alveolar ridges following osseodensification as compared to ridge splitting with simultaneous implant placement using CBCT.

Interventions:

I. Pre-operative phase:

Clinical Examination:

1. Visual examination, palpation and inspection of the entire oral and Para-oral tissues.
2. Preoperative alginate impressions for both the maxillary and the mandibular Ridges.
3. Full mouth scaling and root planing, followed by oral hygiene instructions.
4. The Bucco-Lingual/Palatal alveolar ridge width measurement at site of interest using a bone caliper.
5. Study casts will be made in order to properly evaluate the inter-arch space, occlusion type and direction of forces in regard to the site of the future implant.

Radiographic Examination:

1. A panoramic radiograph for screening purposes:

   * Estimating the residual bone height.
   * Verify the absence of any pathology in the bone.
2. Cone beam computed Tomography (CBCT) for Diagnostic purposes:

   * Detect the Bucco-lingual/palatal alveolar ridge width and height at the site of interest.
   * Detect approximation to any anatomical boundaries (e.g.mental foramen, maxillary sinus floor.)
   * Detect bone type.

II. Surgical phase:

All procedures will be done under strictly aseptic conditions

1. Patients will be anesthetized at the surgical site by the appropriate method using Articaine Hydrochloride 4%.
2. At the site a horizontal incision will be created, extending the entire length of the edentulous area, extending one tooth mesial and distal. Anterior and/or posterior vertical releasing incision will be made as needed.
3. Full thickness mucoperiosteal flap will be raised with complete exposure of the alveolar bone.
4. Bone width will be reconfirmed intrasurgically using a bone caliper. Measurements will be taken at around 1 mm below the crestal margin, to the nearest 0.5mm. Alveolar ridge width measurements will be repeated at second stage surgery.
5. A.For the intervention:

   1. Drilling of bone will commence using the Pilot Drill to the desired depth (Drill speed 800-1500 rpm with copious irrigation).
   2. Osseodensification drilling will begin with the narrowest Densah Bur. (Counterclockwise drill speed 800-1500 rpm with copious irrigation). If when running the bur into the osteotomy a feeling of haptic feedback of pushing up and out of the osteotomy, repetitively lifting off and reapplying pressure with a pumping motion will be applied until the desired depth is reached.
   3. Densah Burs will be used sequentially in small increments. As the bur diameter increases, the bone will slowly expand to the final diameter.
   4. The osteotomy final preparation diameter would be an average diameter that measures 0.5-0.8 mm smaller than the implant average diameter in soft bone, and In hard bone, diameter that measures 0.2-0.5 mm smaller than the implant average diameter.
   5. Implant placement using the drill motor initially, then Finishing placement of the implant to depth with a torque-indicating wrench.
   6. If < 1mm of buccal bone thickness has resulted after osseodensification, bone grafting post implant placement and complete implant coverage will be considered

5.B.For the control:

1. A bone crestal incision will be created, using the piezo-electric surgical tips. The cut will be done through the cortical bone to reach the trabecular bone.
2. One/two vertical cuts will be created by piezo-drill as needed connecting, to the crestal cut.
3. Conventional Drills will be used for osteotomy preparation by wedging it between the two plates of bone.
4. The implant with the proper length and diameter will be gradually engaged to separate the buccal and Lingual/palatal bone until full seating is achieved.

   6. Cover screws will be placed on the implants. 7.Closure of the flap will be done by interrupted sutures using 4-0 resorbable suture materials.

   III. Post-operative phase:

   Post-operative instructions and medication:

   Patient is recommended to:
   1. Maintain a soft diet to avoid trauma to the surgical site.
   2. Place a cold compress superficially on the skin overlying the surgical site immediately. Apply for 30 minutes, then off for 20-30 minutes. This should be done on a near continuous basis (or as much as possible) for the first 48 hours.
   3. Maintain Oral hygiene but avoid surgical site for the first 4 days after surgery.
   4. Medications (Ferrigno et al. 2005)( Garcez-Filho et al.2015) • Augmentin* (1g tablets) will be prescribed twice daily for 5 days to avoid possibility of infection.

      • Ibuprofen** 600mg four times daily for one week.

      • Voltarene*** (75 mg injection I.M.) will be used in case of severe pain, as a rescue.

      • Hexitol**** 0.12% chlorhexidine mouth rinse for 2 weeks.
   5. Sutures will be removed after 2 weeks
   6. Final restoration will be completed after 6 months

      * Augmentin 1g. Medical union pharmaceuticals co. Abu Sultan, Ismailia, Egypt. **BRUFEN 600 (Ibuprofen 600 mg). Kahira Pharm. & Chem. Ind. Co., Under licence from: Abbott Laboratories.

        * Voltarene® 75mg/3ml (IM). Diclofenac natrium. NOVARTIS PHARMA. S.A.E.

          * Hexitol Chlorhexidine Hcl 125 mg / 100 ml. Arab Drug Company (ADCO).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least one missing tooth in need of replacement.
2. Patients having a Bucco-lingual/palatal width of the edentulous alveolar ridge less than 6 mm with a minimum of 3mm residual bone width.
3. Patients having at least 11 mm residual bone height at the proposed edentulous area.
4. The recipient bed of the implant should be free from any pathological conditions.
5. No history of diagnosed bone disease or medication known to affect bone metabolism.
6. Patients who are cooperative, motivated, and hygiene conscious.

Exclusion Criteria:

1. Patients incapable to undergoing minor oral surgical procedures.
2. Patients with insufficient vertical inter-arch space, upon centric occlusion, to accommodate the available restorative components.
3. Patients who have any systemic condition that may contraindicate implant therapy.
4. Patients with modifying habits affecting osteointegration for example, smoking and alcoholism.
5. Patients with parafunctional habits that can overload the implant, such as bruxism and clenching.
6. Patients with impractical expectations about the esthetic outcome of implant therapy.
7. Patients in the growth stage with mixed dentition.
8. Patients with a history of drug abuse.
9. Patients with a history of psychiatric disorder.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-30 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change in bone width | Baseline and six month post surgically
  Using Cone beam computed tomography bone width gain will be reported in millimeters.

SECONDARY OUTCOMES:
Change in Implant stability Quotients | at the time of surgery and 6 month post surgical
  using the Periotest, the implant stability's as an Assessment of osseointegration of dental implants will be reported numerically.Periotest value range -8 to +50. from -8 to 0;Good osseointegration; the implant is well integrated and can be loaded. from+10 to +50;Osseointegration is insufficient; the implant must not be loaded.
soft tissue healing at 1 week using the Healing index by Landry,Turnbull and Howley (1988) to describe the extent of clinical healing after periodontal surgery. | 1 week post surgically.
  Assessed numerically using Healing index by Landry,Turnbull and Howley 1988.The Healing index scores healing with a 5-level score index evaluated with the following parameters: tissue color,presence of granulation tissue, bleeding
  ,suppuration and epithelialisation. by applying a dichotomic scoring system (0/1) with a total score of 5: presence/absence of redness; presence/absence of granulation tissue; presence/absence of suppuration; degree of tissue epithelialization (partial/complete); presence/absence of bleeding.A score range of 1 to 5 is given, with 1 associated with very poor healing and 5 being excellent healing.
soft tissue healing at 2 weeks using the Healing index by Landry,Turnbull and Howley 1988 to describe the extent of clinical healing after periodontal surgery. | 2 weeks post surgically
  Assessed numerically using Healing index by Landry,Turnbull and Howley 1988.The Healing index scores healing with a 5-level score index evaluated with the following parameters: tissue color,presence of granulation tissue, bleeding
  ,suppuration and epithelialisation. by applying a dichotomic scoring system (0/1) with a total score of 5: presence/absence of redness; presence/absence of granulation tissue; presence/absence of suppuration; degree of tissue epithelialization (partial/complete); presence/absence of bleeding.A score range of 1 to 5 is given, with 1 associated with very poor healing and 5 being excellent healing.
Changes in Crestal Bone level | at the time of enrollment and 6 month post surgically
  using the Cone beam computed tomography crestal bone level differences will be evaluated and reported in millimeters.
Pain scale using the numerical Visual analog scale. | 1 week post surgically
  Using the numerical Visual analog scale. Pain sensation will be evaluated and reported. The visual analog scale is a continuous scale made of a horizontal line, about 10 centimeters (100 mm) in length, anchored by 2 extremes descriptors,"no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100).

CONTACTS AND LOCATIONS:
Overall Officials: Radwa A ElMaghrabi, BSC, Principal Investigator — Cairo University; Amr zahran, PHD, Study Director — Cairo University; Ahmed Al barbary, PHD, Study Chair — Cairo University
Locations (1):
- The Faculty of Dentistry -Cairo University, Cairo, Egypt